CLINICAL TRIAL: NCT05146622
Title: SSW Works: A Virtual Learning Environment for Occupational Skin Cancer Prevention Phase I
Brief Title: Virtual Sun Safe Workplaces Ph I
Acronym: SSW Works
Status: Completed | Type: Observational
Sponsor: Klein Buendel, Inc. (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0333; 1R44CA257778-01A1 (NIH)
Record Dates: First submitted 2021-11-23; First posted 2021-12-07 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Skin Cancer
MeSH Terms: conditions — Skin Neoplasms | interventions — Workplace

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Formative Research: Outdoor workers in the United States.
  Interventions: Behavioral: Workplaces in the World

INTERVENTIONS:
Behavioral: Workplaces in the World — Formative research activities to better understand attitudes and behaviors of outdoor workers with respect to UV safety.
  Other Names: Go Sun Smart at Work 2.0

SUMMARY:
Americans who work outdoors are exposed to an extreme amount of solar ultraviolet radiation over a lifetime that substantially increases their risk for developing skin cancer. In Phase I, the feasibility of a virtual learning environment (VLE) for distributing our effective Sun Safe Workplaces (SSW) intervention to American employers will be established with input from senior managers and Hispanic and African American outdoor workers and development and evaluation of a prototype of the SSW Works VLE. In Phase II, the full SSW Works will be produced and tested for effectiveness at improving outdoor workers' sun protection in a randomized trial enrolling employers nationwide.

DETAILED DESCRIPTION:
Americans who work outdoors are exposed to an extreme amount of solar ultraviolet radiation (UV) over a lifetime that substantially increases their risk for developing skin cancer. Annually, skin cancer is diagnosed in over 3.5 million U.S. adults, melanoma kills nearly 7,000 Americans, and treatment costs at least $8 billion. The U.S. Surgeon General has identified occupational sun safety as a national priority. Our team has spent the past two decades developing a successful comprehensive approach to occupational sun protection in 5 trials funded largely by the National Cancer Institute. Sun Safe Workplaces (SSW) combines policy and education to increase workplace actions on sun safety and employee sun protection practices. In this SBIR Fast-Track application, we will develop a virtual learning environment (VLE), SSW Works, to distribute the SSW program to American workplaces. It will be comprised of a database, content management (interactive toolbox), and media platform (trackable training) that tailors the SSW program to management's readiness to innovate on sun safety based Diffusion of Innovations Theory. SSW Works will better integrate SSW into safety training by improving appropriateness for Hispanic and African American workers and conforming with the latest learning management systems technology (LMS). Strong scientific premise comes from the published literature and our 5 previous studies that demonstrated SSW is feasible and effective in public works, public safety, and outdoor recreation workplaces. The Phase I specific aims will establish the feasibility of SSW Works by 1) creating and validating an algorithm to tailor resources and implementation strategies to employers' stages in the diffusion of innovations process; 2) identifying unique attitudes, barriers, and practices related to sun safety among Hispanic and African American employees in focus group discussion and adjusting the SSW content; and 3) creating a prototype of the SSW Works VLE, including inputs, staging algorithm and tailored report, employee training compatible with a popular LMS, and storyboards of brief videos for managers and employees and testing it for feasibility and usability with managers and Hispanic and African American outdoor workers, and confirming that the training can operate within a popular LMS. In Phase II, SSW Works will be fully programmed and tested for effectiveness by achieving the specific aims of: 1) producing the full SSW Works, in English and Spanish, for distribution of the evidence-based SSW and 2) conducting a randomized controlled trial with 20 workplaces evaluating impact of SSW distributed over the SSW Works on employees' sun safety practices (primary outcome). The primary hypothesis is: compared to employers in the minimal information control group, employers assigned to receive SSW Works will have employees that practice more sun protection at posttest. The SBIR Fast-Track research is significant and innovative. SSW Works will have high impact and commercial potential because outdoor workforce is large and at very high risk for skin cancer, improving sun safety will reduce health care costs and save lives, and there are few commercial competitors.

ELIGIBILITY:
Inclusion Criteria:

* Employed part-/full-time at a participating employer
* Work at least 5 hours outdoors per week
* Read English or Spanish
* Complete the pretest survey
* Employed in a management/supervisory position
* Responsible for worksite safety/health policy or education
* Consent to participate

Exclusion Criteria:

* Work exclusively indoors
* Can read neither English nor Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Outdoor workers in the United States.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2021-10-28 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Formative Research Activities | Baseline Only
  Focus Groups and Semi-structured Interviews

CONTACTS AND LOCATIONS:
Overall Officials: Mary Buller, MA, Principal Investigator — Klein Buendel, Inc.
Locations (1):
- Klein Buendel, Inc., Golden, Colorado, United States